CLINICAL TRIAL: NCT02643537
Title: Associated Pathologies Following Luxatio Erecta Humeri: A Retrospective Analysis of 31 Cases and Diagnostic Algorithm
Status: Completed | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Julian Joestl, MD, Medical University of Vienna
Other Study IDs: 2009
Record Dates: First submitted 2015-12-19; First posted 2015-12-31 (Estimated); Last update posted 2015-12-31 (Estimated); Status verified 2015-12

CONDITIONS: Shoulder Dislocation
MeSH Terms: conditions — Shoulder Dislocation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Luxation erecta: All patients with Inferior shoulder dislocation in fixed abduction, also known as luxatio erecta humeri (LEH)

SUMMARY:
The aim of this study was to evaluate the clinical outcome of this rare injury with special emphasis on associated pathologies. Additionally, we aimed to develop an algorithm for the diagnosis of associated pathologies following LEH.

ELIGIBILITY:
Inclusion Criteria:

* Included for analysis were all patients over 18 years of age who have been treated for LEH between at our department.

Exclusion Criteria:

* Only injuries of the affected shoulder were taken into account, non-shoulder related pathologies were not addressed.
* Other types of shoulder dislocation except Luxatio erecta

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Included for analysis were thirty-one patients (11 females (average age 68.2 years) and 20 males (average age 48.3 years)) who have been treated for Laxation erecta between 1992 and 2015.
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 1992-01; Primary Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Functional clinical outcome | at least 2months
  Functional outcome (Range of Motion of the shoulder)

SECONDARY OUTCOMES:
ASSOCIATED PATHOLOGIES | at least 2 months
  Number of participants with associated pathologies (for example fractures of the greater tuberosity, injuries of the rotator cuff or nerve palsy, e.g.) that were connected with this rare injury
Pain | at least 2 months
  Assessment for pain after operative/conservative therapy with the Visual Analog Score for pain